CLINICAL TRIAL: NCT06128746
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Spasticity in Children With Hemiplegic Cerebral Palsy/ Hemiplegia Due to Acquired Brain Injury - a Randomized Controlled Trial
Brief Title: rTMS Treatment of Spasticity in Children With Cerebral Palsy/ Hemiplegia Due to ABI - a RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie Wan Yee Tso (Dr), Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rTMSCPHKU
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: CP (Cerebral Palsy)
Keywords: TMS; Cerebral palsy; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional rTMS group (Experimental): The intervention group will receive 1 Hz active rTMS during treatment, lasting for 20 minutes, follow up by 30 minutes of intensive limb training.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS group (Sham Comparator): The sham group will not receive any Hz of rTMS during treatment, also lasting for 20 minutes with 30 minutes of intensive limb training afterwards.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — 1 Hz rTMS treatment for 20 mins, follow by 30 mins intensive limb training
  Arms: Interventional rTMS group
Device: Sham Repetitive Transcranial Magnetic Stimulation — Sham Hz rTMS treatment for 20 mins, follow by 30 mins intensive limb training
  Arms: Sham rTMS group

SUMMARY:
This RCT aims to investigate the effect of repetitive transcranial magnatic stimulation (rTMS) in treating children with hemiplegoc cerebral palsy. The study will measure any improvement in spasticity after using contra-lesional inhibitory rTMS follow by intensive limb training.

Participants will attend a 10-day rTMS treatment sessions, follow by intensive training of the impaired limb. They will also undergo MRI scans before and after the treatment to investiagte the underlying neurophysiological mechanisms that lead to changes clinically by using TMS as well as MR-DKI. Researchers will compare the intervention group and the sham group to see if rTMS could result in improvement of participants' spasticity.

DETAILED DESCRIPTION:
Cerebral palsy is the most common cause of lifelong physical disability in childhood, with an estimated prevalence of 1.5 per 1000 living biths for primary school-aged children. Spasticity is the most common symptoms in children with cerebral palsy, leading to muscle weakness affecting gross motor functions and causing complications such as pain, contracture and subluzation which will lead to inability to perform activity-based training and subsequently lead to further muscle weakness. Standard therapy with regular physiotherapy and occupational therapy are essential but time-consuming and the effects might not last for longer duration. Patients or caregivers decline medications because of side effects drowsiness while other interventions such as intra-thecal baclofen pump, rhizotomy or surgery are invasive.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that has the ability to modulate excitation of the motor cortex area of the brain. There were past studies suggesting that using contralesional inhibitory rTMS was safe and feasible for patients with paediatric subcortical stroke and seemed to improve hand function in patients with hemiparesis. However, limited studies have been published on the effects of rTMS on improving spasticity in children with cerebral palsy. Hence, the objective of this study is to use low-frequency rTMS to the contra-lesional hemisphere in children with hemiplegic cerebral palsy to investigate if rTMS follow by intensive limb training would improve spasiticity of these children and whether the improvement can be sustained for a longer time. The underlying mechanisms that lead to the changes clinically will also be investigated by TMS and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 7 years and 18 years
* Diagnosis of cerebral palsy with hemiplegia
* Upper limb spasticity ≥ 1
* IQ ≥ 50

Exclusion Criteria:

* Any contra-indications to rTMS
* Severe spasticity (score of 4 or more in Ashworth scale)
* Uncontrollable epilepsy
* History of Botulinum toxin A injection in previous 6 months
* Upper limb casting in previous 6 months

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Day 10, 17 of intervention and 2 months post intervention
  Clinical measure of spasticity. Scores range from 0 to 4, with a higher score indicate worse in muscle tone
The range of motion scores | Day 10, 17 of intervention and 2 months post intervention
  ROM of thumb adduction, wrist dorsal flexion and extension, and elbow dorsal flexion and extension. Patients' range of motion score will be compared to the normative values

SECONDARY OUTCOMES:
Zancolli scale | Day 10, 17 of intervention and 2 months post intervention
  Severity of forearm alignment. Scores range from 0 to 3 with a higher score indicate worse hand function
House functional classification scale | Day 10, 17 of intervention and 2 months post intervention
  Rating of functional use of the impaired upper limb. Scale consists of nine grades from 0 (does not use) to 8 (full spontaneous use)
Gross motor function measure | Day 10, 17 of intervention and 2 months post intervention
  Changes in motor function. A 4-point Likert scale with higher score indicates better motor function
Assisting hand assessment | Day 10, 17 of intervention and 2 months post intervention
  Test of hand function
Pediatric Quality of Life Cerebral Palsy module | Day 10, 17 of intervention and 2 months post intervention
  Quality of life measurement. Scores range from 0 to 100 with higher score indicate better quality of life.
MRI Brain: fMRI and DKI | Day 10, 17 of intervention and 2 months post intervention
  Functional MRI and Diffusion Kurtosis Imaging measuring the brain microstructural changes and structural connectivity during the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Li Ka Shing Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No